CLINICAL TRIAL: NCT03485131
Title: Transcranial Direct-current Stimulation (tDCS) in Treatment Refractory Auditory Hallucinations: A Pilot Study
Brief Title: Transcranial Direct-current Stimulation (tDCS) in Treatment Refractory Auditory Hallucinations
Acronym: tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manhattan Psychiatric Center (Other)
Responsible Party: Principal Investigator, Jean-Pierre Lindenmayer, Director of Research, Manhattan Psychiatric Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1409
Record Dates: First submitted 2016-03-01; First posted 2018-04-02 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Auditory Hallucination; Schizophrenia
MeSH Terms: conditions — Hallucinations; Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Two group randomized, parallel design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Raters were blind as was PI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Transcranial direct-current stimulation (Experimental): Intervention of 2 mAmp Transcranial direct-current stimulation treatments given twice daily for 20 min each per day for 4 weeks on consecutive weekdays. Twice-daily sessions were separated by at least 3 hours (one in the AM and the other one in the PM)
  Interventions: Device: Transcranial direct-current stimulation (tDCS)
- Sham tDCS (Sham Comparator): Intervention of placebo stimulation with ranscranial direct-current stimulation(sham tDCS), the stimulation parameters were displayed, but after 40 seconds of real stimulation of 2 mAmp to simulate the tDCS induced skin sensation, only a small current pulse was delivered every 550 msec (110 mAmp over 15 msec) through the remainder of the 20-minute period
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Transcranial direct-current stimulation (tDCS) — Stimulation sessions will be conducted twice a day on 5 consecutive weekdays. The twice daily sessions will be separated by at least 3 hours (one in the morning and the other one in the PM). The duration of treatment will be 4 weeks
  Other Names: Active Transcranial direct-current stimulation (tDCS)'
  Arms: Transcranial direct-current stimulation
Device: Placebo — Placebo/sham stimulation: After 40 seconds of real stimulation of 2 mAmp to simulate the tDCS induced skin sensation, only a small current pulse is delivered every 550 msec (110 mAmp over 15 msec) through the remainder of the 20-minute period
  Other Names: Sham Transcranial direct-current stimulation (tDCS)
  Arms: Sham tDCS

SUMMARY:
This is a 4 week therapeutic pilot study with a 4 week follow-up period involving inpatients with treatment resistant DSM-IV schizophrenia or schizoaffective disorder diagnosis. Each eligible subject will receive either 20 minutes of active tDCS (transcranial direct-current stimulation) or sham stimulation twice a day on 5 consecutive weekdays for 4 weeks with a 4 week follow-up period.

DETAILED DESCRIPTION:
The aim in this study is to conduct a pilot study on the efficacy of tDCS by assessing its efficacy in treatment refractory auditory verbal hallucinations in inpatients with chronic schizophrenia. Based on and expanding the findings by Brunelin et al. the hypothesis is that tDCS treatment with the cathode on the left temporal-parietal junction and the anode on the left dorsolateral prefrontal cortex can reduce the severity of auditory verbal hallucinations in patients with treatment refractory schizophrenia. The impact of tDCS on other schizophrenia symptoms in secondary exploratory outcome analyses together with the examination of the durability of an ameliorating effect will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient adults (age 18-65 years) who meet diagnostic criteria for schizophrenia or schizoaffective disorder (using the Structured Clinical Interview for DSM)
* Auditory hallucinations without remission over 5 years (remission is defined as a period of 4 weeks without hallucinations) as documented in the patients' medical record
* Failure to respond to two previous adequate antipsychotic trials with adequate duration and adequate dosage
* Screening PANSS total rating of > 70
* PANSS hallucinatory behavior item > 4
* Capacity and willingness to sign informed consent
* On a stable antipsychotic regimen 4 weeks prior to screening and for the duration of the trial
* Normal hearing
* If female and not infertile, must agree to use one of the following forms of contraception for the duration of study participation: systemic hormonal treatment, an interuterine device (IUD) which was implanted at least 2 months prior to screening, or "double-barrier" contraception
* Willing to wear the tDCS device.

Exclusion Criteria:

* Prior history of seizure, other than that induced by Electro Convulsive Therapy
* Family history of seizures
* Significant unstable medical condition
* Pregnancy or women of childbearing capacity not using a medically accepted form of contraception when engaged in sexual intercourse
* Inability to provide informed consent
* Actively suicidal and or showing violent behavior
* Significant organic brain pathology by history and neurological examination, inclusive of history of head trauma, loss of consciousness for more than 5 minutes; intracranial metal implants, known structural brain lesion, devices that may be affected by transcranial Direct Current Stimulation (tDCS) (pacemaker, medication pump, cochlear implant, implanted brain stimulator)
* Active substance abuse
* Increased intracranial pressure, unstable cardiovascular disease, sleep apnea
* Individuals with a clinically defined neurological disorder
* Frequent and persistent migraines
* History of adverse reaction to neurostimulation or open skin wounds that would preclude safe placement of tDCS electrodes
* Current use of medications known to lower seizure threshold (serotonergic or tricyclic antidepressants)
* If pregnant or breast feeding at the time of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Reduction on the severity of auditory verbal hallucinations | 8 weeks
  Reduction of Auditory Hallucinations Rating Scale (AHRS (12) items)

SECONDARY OUTCOMES:
Impact of tDCS on other schizophrenia symptoms | 8 weeks
  Reduction of scores in Positive and Negative Symptom Scale
Impact of tDCS on Clinical Global Impression | 8 weeks
  Global Severity of Illness measure
Impact of tDCS on MATRICS | 8 weeks
  MATRICS: Comprehensive assessment of cognitive functions

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Lindenmayer, MD, Principal Investigator — Manhattan Psychiatric Center
Locations (1):
- Manhattan Psychiatric Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nitsche MA, Boggio PS, Fregni F, Pascual-Leone A. Treatment of depression with transcranial direct current stimulation (tDCS): a review. Exp Neurol. 2009 Sep;219(1):14-9. doi: 10.1016/j.expneurol.2009.03.038. Epub 2009 Apr 5. PMID 19348793